CLINICAL TRIAL: NCT00916708
Title: Appropriateness Evaluation of Follow up Procedures in Gynaecology Oncology TOTEM Study: Multicentric Randomized Controlled Clinical Trial Between Two Follow up Regimens With Different Tests Intensity in Endometrial Cancer Treated Patients.
Brief Title: Trial Between Two Follow up Regimens With Different Test Intensity in Endometrial Cancer Treated Patients
Acronym: TOTEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other); Rete Oncologica Piemonte, Valle d'Aosta (Other)
Responsible Party: Principal Investigator, Paolo Zola, Paolo Zola MD, Study Coordinator, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TOTEM
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; follow up; relapse
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive follow up (Experimental): Intensive follow up in low-risk patients Intensive follow up in high-risk patients
  Interventions: Procedure: Intensive/Low-Risk follow up (IA G1; IA G2); Procedure: Intensive/High-Risk follow up (≥ IA G3)
- Minimalist follow up (Experimental): Minimalist follow up in low-risk patients Minimalist follow up in high-risk patients
  Interventions: Procedure: Minimalist/Low-Risk follow up (IA G1; IA G2); Procedure: Minimalist/High-Risk follow up (≥ IA G3)

INTERVENTIONS:
Procedure: Intensive/Low-Risk follow up (IA G1; IA G2) — - First 2 years of FU since the end of primary treatment: clinical visit* every 4 months; Pap tests; chest, abdomen, pelvis CT every 12 months
  - Since the third to the fifth year of FU: clinical visit* every 6 months; Pap test every 12 months
  * clinical visit with gynecological exploration
  Arms: Intensive follow up
Procedure: Intensive/High-Risk follow up (≥ IA G3) — - First 3 years of FU since the end of primary treatment: clinical visit*, Ca125, trans-vaginal and abdominal ultrasound every 4 months (except in conjunction with TC); Pap smear, abdomen, pelvis CT every 12 months
  - In the fourth and fifth years of FU: clinical visit*, Ca125, trans-vaginal and abdominal ultrasound every 6 months (except in conjunction with TC) Pap smear; chest, abdomen, pelvis CT every 12 months
  * clinical visit with gynecological exploration
  Arms: Intensive follow up
Procedure: Minimalist/Low-Risk follow up (IA G1; IA G2) — - First 5 years of FU since the end of primary treatment: clinical visit* every 6 months.
  * clinical visit with gynecological exploration
  Arms: Minimalist follow up
Procedure: Minimalist/High-Risk follow up (≥ IA G3) — - First 2 years of FU since the end of primary treatment: clinical visit* every 4 months; chest, abdomen, pelvis CT every 12 months
  - Since the third to the fifth year of surveillance: clinical visit* every 6 months.
  * clinical visit with gynecological exploration
  Arms: Minimalist follow up

SUMMARY:
This study aims to compare two different follow up regimens with different test intensity in endometrial cancer treated patients.

If eligibility criteria are satisfied and the written informed consensus is obtained, patients are stratified inside the centre according to their risk level:

* Group 1 : patients at low risk of recurrence [stage IA G1 and stage IA G2]
* Group 2 : patients at high-risk of recurrence [≥ stage IA G3] (Ethics Committee amendment of 14th September 2010, use new 2010 FIGO classification for endometrial cancer!)

In each group patients will be randomized in two regimens of follow up:

1. Minimalist (Arm 1)
2. Intensive (Arm 2)

Features of each arm are listed in "Arms" item.

DETAILED DESCRIPTION:
The procedure for centralized randomization, with blocks of variable length, will take place within each layer with 1:1 ratio and will be implemented within the centralized database, with sequences generated by dedicated software. The recruitment and randomization has to be registered on the website (www.epiclin.cpo.it) no later than 20 days after histological examination has been received. If patients do not need any kind of adjuvant therapy they will start follow-up program according to the regimen chosen for them at randomization, if adjuvant therapy is needed the patient at first will be registered and the randomization will be deferred at the end of treatment.

In presence of symptoms or signs detected during the clinical visit which may suppose a recurrence or in presence of abnormal tests, the clinician has to prescribe all medical tests and examinations required. The tests carried out in addition to follow-up scheduled program must be reported in the database. Nevertheless patients continue to be followed for the assessment of the performance status at 5 years, but the follow-up schedule is up to the clinician. An interim analysis is scheduled in 3.5 years starting from the beginning of recruitment (based on approximately 1 / 3 of the total expected events, when about 4 / 5 cases have already been enrolled). Patients will be stratified by recruitment Center, by level of risk (calculated according to the stage of the disease, the histotype and the grading) and by type of treatment performed.

The focus of the study is to:

* Compare the effect of two FU regimens on 5-years OS
* Evaluate the difference in diagnosis anticipation
* Evaluate the difference in terms of recurrences
* Describe the compliance and QoL of patients
* Evaluate the cost-effectiveness and the cost-utility

ELIGIBILITY:
Inclusion Criteria:

* patients treated surgically for endometrial cancer, if in complete clinical remission confirmed by imaging stage FIGO I-IV
* no previous or concurrent neoplasia (with the exception of carcinoma in situ of the cervix and basalioma of the skin)
* other contemporaneous RCT may be allowed if there is not any restriction concerning follow up
* obtaining a written informed consensus before randomization
* age > 18 years

Exclusion Criteria:

* presence of any psychological, familial, sociological or geographical condition that could potentially limit the compliance to the protocol and the follow-up planned: all these situations must be discussed with the patient before the randomization
* previous, concurrent or second malignancies endometrial carcinoma in the context of a hereditary syndrome
* conditions which contraindicate medical tests scheduled according to follow-up regimen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1884 (Actual)
Dates: Start 2008-09; Primary Completion 2018-07-31 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Seven years

SECONDARY OUTCOMES:
Progression-free survival | Seven years
Proportion of complications, second cancers, co-morbidity | Seven years
Proportion of asymptomatic patients with diagnosis of relapse | Seven years
Proportion of subjects who complete the two different regimes follow up | Seven years

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Zola, MD, Principal Investigator — Azienda Ospedaliera Città della Salute e della Scienza di Torino - University of Turin
Locations (1):
- Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gadducci A, Fuso L, Cosio S, Landoni F, Maggino T, Perotto S, Sartori E, Testa A, Galletto L, Zola P. Are surveillance procedures of clinical benefit for patients treated for ovarian cancer?: A retrospective Italian multicentric study. Int J Gynecol Cancer. 2009 Apr;19(3):367-74. doi: 10.1111/IGC.0b013e3181a1cc02. PMID 19407561
- [Background] Zanagnolo V, Minig LA, Gadducci A, Maggino T, Sartori E, Zola P, Landoni F. Surveillance procedures for patients for cervical carcinoma: a review of the literature. Int J Gynecol Cancer. 2009 Apr;19(3):306-13. doi: 10.1111/IGC.0b013e3181a130f3. PMID 19407551
- [Background] Zola P, Fuso L, Mazzola S, Piovano E, Perotto S, Gadducci A, Galletto L, Landoni F, Maggino T, Raspagliesi F, Sartori E, Scambia G. Could follow-up different modalities play a role in asymptomatic cervical cancer relapses diagnosis? An Italian multicenter retrospective analysis. Gynecol Oncol. 2007 Oct;107(1 Suppl 1):S150-4. doi: 10.1016/j.ygyno.2007.07.028. Epub 2007 Sep 14. PMID 17868785
- [Background] Zola P, Fuso L, Mazzola S, Gadducci A, Landoni F, Maggino T, Sartori E. Follow-up strategies in gynecological oncology: searching appropriateness. Int J Gynecol Cancer. 2007 Nov-Dec;17(6):1186-93. doi: 10.1111/j.1525-1438.2007.00943.x. Epub 2007 Apr 26. PMID 17466042
- [Background] Gadducci A, Cosio S, Zola P, Landoni F, Maggino T, Sartori E. Surveillance procedures for patients treated for epithelial ovarian cancer: a review of the literature. Int J Gynecol Cancer. 2007 Jan-Feb;17(1):21-31. doi: 10.1111/j.1525-1438.2007.00826.x. PMID 17291227
- [Derived] Rosato R, Ferrero A, Mosconi P, Ciccone G, Di Cuonzo D, Evangelista A, Fuso L, Piovano E, Pagano E, Laudani ME, Pace L, Zola P; TOTEM Collaborative Group. Impact of different follow-up regimens on health-related quality of life and costs in endometrial cancer patients: Results from the TOTEM randomized trial. Gynecol Oncol. 2024 May;184:150-159. doi: 10.1016/j.ygyno.2024.01.050. Epub 2024 Feb 3. PMID 38309033
- [Derived] Zola P, Ciccone G, Piovano E, Fuso L, Di Cuonzo D, Castiglione A, Pagano E, Peirano E, Landoni F, Sartori E, Narducci F, Bertetto O, Ferrero A; TOTEM Collaborative Group. Effectiveness of Intensive Versus Minimalist Follow-Up Regimen on Survival in Patients With Endometrial Cancer (TOTEM Study): A Randomized, Pragmatic, Parallel Group, Multicenter Trial. J Clin Oncol. 2022 Nov 20;40(33):3817-3827. doi: 10.1200/JCO.22.00471. Epub 2022 Jul 20. PMID 35858170
- See also: The recruitment of patients has to be registered on the website (http://www.epiclin.it). On the website patients are randomized and crf are available to register follow up appointment — http://www.epiclin.it